CLINICAL TRIAL: NCT02033135
Title: Paclitaxel Eluting Stent or Exercise for Thigh Atherosclerosis (PESETA)
Brief Title: Paclitaxel Eluting Stent or Exercise for Thigh Atherosclerosis
Acronym: PESETA
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Lise Pyndt Jørgensen, MD, Ph. D. student, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H 4 2012 027
Record Dates: First submitted 2014-01-08; First posted 2014-01-10 (Estimated); Last update posted 2014-01-10 (Estimated); Status verified 2014-01

CONDITIONS: Peripheral Arterial Disease
Keywords: Atherosclerosis; Intermittent claudication; Angioplasty
MeSH Terms: conditions — Peripheral Arterial Disease; Atherosclerosis; Intermittent Claudication | interventions — Angioplasty

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Angioplasty with Zilver PTX (Experimental): Angioplasty and stenting with a polymer free paclitaxel-eluting stent (Zilver-PTX) plus unsupervised exercise therapy, smoking cessation advice and best medical therapy.
  Interventions: Procedure: Angioplasty with Zilver PTX; Other: Best medical treatment; Device: Zilver PTX
- Best medical treatment (Active Comparator): Unsupervised exercise therapy, smoking cessation advice and best medical therapy.
  Interventions: Other: Best medical treatment

INTERVENTIONS:
Procedure: Angioplasty with Zilver PTX — Angioplasty and stenting with a polymer free paclitaxel-eluting stent (Zilver-PTX)
  Arms: Angioplasty with Zilver PTX
Other: Best medical treatment — Treatment with antiplatelet and statins, smoking cessation advice and unsupervised walking exercise.
Device: Zilver PTX
  Arms: Angioplasty with Zilver PTX

SUMMARY:
This randomized clinical study is intended to evaluate the use of Zilver PTX stents for treatment of thigh atherosclerosis.

Research question: Is there an adjuvant benefit of angioplasty and stenting using the new paclitaxel eluting stent, Zilver-PTX, over risk factor modification and medical therapy alone in patients with stable, mild to moderate intermittent claudication caused by femoropopliteal lesions suitable for endovascular management.

ELIGIBILITY:
Inclusion Criteria:

* Patient has signed and dated the informed consent.
* Patient has 1- 2 documented stenotic or occluded atherosclerotic lesions (up to 18 cm long) of the above-the-knee femoropopliteal artery, that meet all of the inclusion criteria and none of the exclusion criteria.
* Reference vessel (the above-the-knee femoropopliteal artery) diameter of 4 mm to 9 mm.
* Taget lesion(s) should be accessible for stenting, as imaged with angiography (digital subtraction, MRI or CTI), i.e. proximal cm of SFA must be open
* Patient has a de novo or restenotic lesion(s) with >50% stenosis documented angiographically and no prior stent in the target lesion.
* Patient has symptoms of peripheral arterial disease classified as Rutherford Category 2 (moderate claudication) or 3 (severe claudication) lasting for at least 3 months. (Positive Claudication Questionnaire)
* Exercise therapy, smoking cessation advise and best medical therapy must have been implemented at least 3 months ago and without significant clinical effect.
* Patient has a resting ABI <0.9 or an abnormal exercise ABI (decrease of more than 0.15) if resting ABI is normal. Patient with incompressible arteries (ABI >1.2) must have a TBI <0.8.
* Patient agrees to return for a clinical status assessment and duplex ultrasound at 6 weeks, 6 months, 12 months, and at 24 months.

Exclusion Criteria:

* Patient is pregnant, breast-feeding or under 18 years of age.
* Patient unable to understand and sign informed consent forms
* Patient is simultaneously participating in another investigational drug or device study.
* Patient has any planned surgical or interventional procedure within 30 days after the study procedure.
* Patient in whom antiplatelet and/or anticoagulant therapy is contraindicated.
* Patient has known hypersensitivity or contraindication to aspirin, antiplatelet medication, contrast dye, paclitaxel or nitinol.
* Patient 2-3 patent crural vessel runoff with <50% stenosis throughout its course.
* Activity limited by co-morbid condition other than claudication, for example: severe coronary artery disease; angina pectoris; chronic lung disease; neurological disorder such as hemiparesis; arthritis, or other musculoskeletal conditions including amputation and BMI > 40
* Other active significant medical problems such as cancer, known chronic renal disease (serum creatinine greater than 2.0 mg/dl within 60 days or renal replacement therapy), known chronic liver disease or anaemia, active substance abuse, or known history of dementia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2012-06; Primary Completion 2015-04 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
Maximal walking distance | 24 months
  Walking distance will be quantified by standardized treadmill testing using constant speed of 3 km per hour with no incline for a maximum of 5 minutes.

SECONDARY OUTCOMES:
Ankle brachial pressure indices | 24 months
  a measure of the peripheral bloodpressure
Quality of life | 24 months
  Quality of life is evaluated by using questionnaires
Cost of the treatment | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Torben V Schroeder, MD, MDSc, Study Director — Dept. of Vasc. Surg., Rigshospitalet, Blegdamsvej 9, 2100 KBH Ø, Denmark
Locations (1):
- Rigshospitalet, Copenhagen, Østerbro, Denmark